CLINICAL TRIAL: NCT05714826
Title: Comprehensive Optimization At-time of Radical Cystectomy Intervention Through Peri-operative Patient Care Program
Brief Title: Comprehensive Optimization At-time of Radical Cystectomy Intervention
Acronym: COARC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, yair lotan, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU-2022-1221
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Bladder Cancer; Radical Cystectomy
Keywords: Peri-operative
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: It is a prospective randomized study that implements a multi-modal digitally based comprehensive health optimization program in the pre and post-operative setting in patients undergoing radical cystectomy for muscle invasive bladder cancer. Two patient groups will be enrolled and randomized where one group will go through the peri-operative optimization programs and the other group will receive the usual pre-op care followed by post-op care via standard follow-up protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Preop intervention Arm Referral to Perioperative Optimization of Senior Health (POSH) Program Remote patient monitoring device orientation, initial intake, and education UTSW ERAS protocol perioperatively Inpatient geriatrics co-management Monitored recovery Post-operative monitoring with Acticare for 90 days Post-op specialist continuity of care
  Interventions: Other: Preop Intervention and Monitored Recovery
- Control Arm (Active Comparator): Enhanced Recovery After Surgery Usual referral and recovery care as needed Standard follow-up protocol
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Preop Intervention and Monitored Recovery — Perioperative Optimization of Senior Health (POSH) Program; patient monitoring by device orientation, initial intake, education; ERAS protocol, inpatient geriatric co-management; and remote monitoring with Acticare device; post-op continuity of care
  Other Names: Monitored recovery during post-operative phase
  Arms: Intervention Arm
Other: Usual Care — ERAS, Usual referral and recovery care, and Standard follow-up protocol
  Arms: Control Arm

SUMMARY:
The proposed study is aimed at a comprehensive optimization at-time of radical cystectomy (COARC) intervention that focuses on patient optimization throughout the perioperative continuum, from the pre-operative setting to the post-operative period, among patients undergoing radical cystectomy for bladder cancer. This multi-modal strategy will focus on three phases of care around surgery: the pre-operative, peri-operative, and post-operative phases. The intervention group will focus on multiple areas of patient optimization including remote patient monitoring for the earlier identification of potential complications. The overall study mission is to decrease complication rates after radical cystectomy using this comprehensive approach.

DETAILED DESCRIPTION:
The proposed study includes the following-

Part I: Pre-operative period After randomization, patients in the intervention group will be referred to the Perioperative Optimization of Senior Health (POSH) program where they will undergo nutritional, functional, and global health assessment. The POSH team will refer patients as indicated to nutrition, physical medicine and rehabilitation, and other consultants to optimize their preoperative fitness for surgery.

Patients in the intervention group will also receive a Remote Patient Monitoring (RPM) Ipad from ActiCare Health, which will serve as their remote monitoring device and educational tool. At enrollment, they will be asked to complete an initial steps intake using a pedometer that will be provided to them. They will be asked to input vital signs once per week after receiving the Ipad to become familiar with the platform pre-operatively.

At enrollment, patients in both groups will also be asked to complete a patient reported Bladder Cancer Index questionnaire, a survey that tracks quality of life in patients with bladder cancer.

Part II: Perioperative period Both the intervention and control groups will undergo standard of care Enhanced Recover After Surgery (ERAS) bladder cancer protocol, which is a medication and peri-operative management protocol developed by the anesthesia and urology departments specifically for bladder cancer patients undergoing radical cystectomy.

While admitted in the hospital recovering from surgery, patients in the intervention group will automatically receive co-management from the POSH team.

Part III: Post-operative period Both the intervention and the control groups will be followed for 90 days post-operatively. The intervention group will use the RPM Ipad to input vital signs, weight, and pedometer steps 3x/week and on an as needed basis over the follow-up period which will be monitored by the ActiCare Health 24/7 clinical support team. Abnormal parameters will be set so that the UT Southwestern Medical Center clinical care team is alerted to any abnormal values.

ELIGIBILITY:
Inclusion Criteria:

* Adults equal to or more than 18 years old
* Diagnosis of bladder cancer with plan to undergo radical cystectomy
* Agrees to participate in study procedures

Exclusion Criteria:

* Patients undergoing cystectomy for diagnosis other than bladder cancer
* Do not provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2026-05-25 (Estimated); Study Completion 2026-08-24 (Estimated)

PRIMARY OUTCOMES:
90 day complication rate | 90 days
  Number of occurrences of complications at 90 days in patients in post-operative phase

SECONDARY OUTCOMES:
30 day complication rate | 30 days
  Number of occurrences of complications at 30 days in patients in post-operative phase
Readmission rates | 90 days
  Number of readmissions
Adherence to the intervention | 90 days
  It is assessed via patient-self report measure
Changes in functional fitness as measured by step count | Baseline, 90 days
  Changes in functional fitness will be measured by step count
QOL changes as measured by the Bladder Cancer Index and FACT-Bl-Cys Questionnaire measures | Baseline, 90 days
  Changes in patient reported outcomes will be measured by QOL (Bladder Cancer Index questionnaire). Possible scores range from 0-100, where higher scores indicate better HRQOL outcome.
  Changes will also be measured using the FACT-Bl-Cys tool to assess changes in bladder related quality of life in patients undergoing cystectomy over the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Lotan, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No